CLINICAL TRIAL: NCT05292404
Title: Impact of Early PCSK9 Inhibitor Treatment on Heart After Acute Myocardium Infarction： a Muti-center, Open-label, Randomized Controlled Trial
Brief Title: Impact of Early PCSK9 Inhibitor Treatment on Heart After Acute Myocardium Infarction
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Tong Ren Hospital (Other)
Collaborators: China Cardiovascular Association (Other)
Responsible Party: Principal Investigator, Hou Lei, Principal Investigator, Shanghai Tong Ren Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ShanghaiTRH-HL2022
Record Dates: First submitted 2022-03-13; First posted 2022-03-23 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-12

CONDITIONS: Acute Myocardial Infarction
MeSH Terms: interventions — alirocumab

STUDY DESIGN:
Intervention Model Description: PCSK9 inhibitor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Early PCSK9 inhibitor treatment group (Experimental)
  Interventions: Drug: alirocumab
- conventional treatment group (Other)
  Interventions: Other: conventional treatment

INTERVENTIONS:
Drug: alirocumab — In the PCSK9 inhibitor group, a dose of PCSK9 inhibitor (alirocumab,75mg) was injected subcutaneously immediately after PPCI and was administered every two weeks thereafter for 3 months
  Arms: Early PCSK9 inhibitor treatment group
Other: conventional treatment — conventional treatment were given according to international uniformguidelines
  Arms: conventional treatment group

SUMMARY:
This is a multi-center, prospective, randomized, controlled study. The patients with STEMI who were to undergo PPCI were divided into PCSK9 inhibitor group (n=80) and conventional treatment group (n=80) using the interactive web response system (IWRS), at a 1:1 ratio. In the PCSK9 inhibitor group, a dose of PCSK9 inhibitor (alirocumab) was injected subcutaneously immediately after PPCI and was administered every two weeks thereafter for 3 months; the control group received conventional treatment. Cardiac Magnetic Resonance Imaging (MRI) were used to measure myocardial salvage index at 1 week after operation as primary endpoints. Eject fraction at 6 months after operation will also be measured by MRI as secondary endpoints. Serum TnI/T，CKMB levels were detected q8h for three times and and LDL-C levels were detected at 1 month, 3 months and 6 months after operation. Blood inflammation indicators were detected before and 1 week after the operation, and 6 months after the operation.

ELIGIBILITY:
Inclusion Criteria:

1. The age is greater than 18 years old and less than or equal to 80 years old.
2. Patients who are clinically diagnosed with STEMI onset within 24 hours and who are planning to undergo PPCI .
3. Signed informed consent.

Exclusion Criteria:

1. Patients who are allergic to PCSK9 inhibitors.
2. Multivessel disease planned for selective intervention within half a year.
3. Patients who have previously undergone revascularization.
4. Pregnant women or women who plan to become pregnant in the next 2 years.
5. Patients whose life expectancy is less than 1 year.
6. Severe liver or kidney dysfunction (ALT>5 times ULA, eGFR<15ml/min/1.73m2)
7. Known active malignant tumor diseases.
8. Patients considered by the investigator to be unsuitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
myocardial salvage index | 1 week after operation
  measured by Magnetic Resonance Imaging (MRI)

SECONDARY OUTCOMES:
Eject fraction | at 6 months after operation
  measured by MRI

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - nineth people's hospital, School of Medicine, shanghai jiaotong university, Shanghai, Shanghai Municipality
  - Shanghai chest hospital, Shanghai, Shanghai Municipality
  - Shanghai tongren hospital, Shanghai, Shanghai Municipality
  - tenth people's hospital, tongji university, Shanghai, Shanghai, Shanghai Municipality
  - Songjiang hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Xia J, Wang X, Zhou J, Wang D, Pang Y, Xu X, Sang Z, Zhang Y, Zhang J, Wu S, Xiao Z, Hou L. Impact of early PCSK9 inhibitor treatment on heart after percutaneous coronary intervention in patients with STEMI: Design and rationale of the PERFECT II trial. Front Cardiovasc Med. 2022 Sep 23;9:1009674. doi: 10.3389/fcvm.2022.1009674. eCollection 2022. PMID 36211588